CLINICAL TRIAL: NCT06812637
Title: Efficacy and Safety of Wharton's Jelly-Derived Mesenchymal Stem Cell Exosomes in the Treatment of Diabetic Foot Ulcers: A Randomized Controlled Trial
Brief Title: Efficacy and Safety of Wharton's Jelly-Derived Mesenchymal Stem Cell Exosomes in the Treatment of Diabetic Foot Ulcers: A Double-blinded Randomized Controlled Clinical Trial
Acronym: WJ-MSC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Abdallah Mohammed Hafez, Assistant lecturer, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WJ-MSC-exo in diabetic foot
Record Dates: First submitted 2025-02-02; First posted 2025-02-06 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Foot Ulcer (DFU); Exosomes
Keywords: Exosomes; Diabetic foot ulcer; WJ-MSC
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This was a prospective, randomized, double-blind, placebo-controlled clinical trial conducted to evaluate the efficacy and safety of WJ-MSC-derived exosomes gel in patients with diabetic foot ulcers (DFUs).
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treated group (Experimental): 40 patients received standard of care (SOC) with Wharton jelly derived mesenchymal stem cell (WJ - MSC) exosome gel once weekly for 4 weeks followed by follow up for 16 weeks
  Interventions: Drug: WJ-MSC- Exosomes; Combination Product: SOC (Standard of care)
- Control group (Other): 35 patients received standard of care (SOC) only for 4 weeks followed by follow-up for 16 weeks.
- Placebo group (Placebo Comparator): 35 patients received received a visually identical saline-based formulation once weekly for 4 weeks followed by follow up for 16 weeks together with SOC

INTERVENTIONS:
Drug: WJ-MSC- Exosomes — warton jelly derived mesenschymal stem cell derived exosomes dissolved in CMC
  Arms: Treated group
Combination Product: SOC (Standard of care) — Wound depridement for necrotic parts , local antibiotic , dressing , unloading
  Arms: Treated group
Other: Vehicle (placebo) — Vehicle for the MSC-EXO

SUMMARY:
Study effeciency and safety of WJ-MSC derived exosomes in DFU healing

DETAILED DESCRIPTION:
Diabetic foot ulcers (DFUs) represent a significant complication of diabetes mellitus, affecting a substantial proportion of patients and often leading to severe morbidity, prolonged hospital stays, and increased healthcare costs [1]. The management of DFUs remains a considerable challenge due to their chronic nature and the complex interplay of factors that impede healing, including poor blood circulation, neuropathy, and infection and this leads to the increase in the number of amputations [2].

The prevalence of diabetes mellitus (DM) is rising globally, with projections of affected individuals increasing from 463 million in 2019 to 642 million by 2040 [3], particularly in regions like the Middle East and North Africa (MENA), where Egypt ranks among the top 10 countries with the highest diabetes prevalence [4].Diabetic foot ulcers (DFUs) are a common and debilitating complication of DM, with a lifetime risk of 19-34% among diabetic patients and accounting for 85% of diabetic lower-limb amputations (DLLA) [5, 6].These ulcers significantly contribute to morbidity, prolonged hospitalizations, and a high socio-economic burden while being associated with post-amputation mortality rates of 24.6% within 5 years and 45.4% within 10 years [7].

The scale of this challenge demands urgent attention to innovative, cost-effective interventions to alleviate both human suffering and financial strain[8], various approaches have been developed to enhance healing and prevent recurrence, such as advanced wound dressings, offloading techniques, and the use of growth factors or skin substitutes [9]. But they are still far from ideal. As such, there is an urgent need for innovative therapeutic strategies that can effectively promote wound healing and improve patient outcomes. applications.

In recent years, mesenchymal stem cell (MSC) - derived exosomes have garnered attention in regenerative medicine. Exosomes are small extracellular vesicles that facilitate intercellular communication by transporting proteins, lipids, and nucleic acids. MSC-derived exosomes have demonstrated the ability to modulate inflammation, promote angiogenesis, and enhance tissue repair across various conditions, including cardiovascular diseases, osteoarthritis, and chronic wounds [10].

Traditionally, bone marrow (BM) has been the primary source of pluripotent MSCs. However, harvesting BM requires an invasive procedure, and with advancing age, the quantity, differentiation potential, and lifespan of BM-derived MSCs decline significantly So alternative sources such as the umbilical cord and adipose tissue (AD) have gained attention [11] . Among these, umbilical cord-derived MSCs, specifically those from Wharton's jelly (WJ), known as Wharton's jelly mesenchymal stem cells (WJ-MSCs) have unique properties. WJ-MSCs are highly accessible, ethically uncontroversial, and offer significant advantages, including a strong differentiation potential and an immunoprivileged status. Moreover, they exhibit characteristics similar to embryonic stem cells including rapid cell division and high expansion capacity[12].

Experimental evidence suggests that WJ-MSCs demonstrate superior proliferation potential compared other MSC such as adipose tissue-derived MSCs (AD-MSCs). These properties position WJ-MSCs as an attractive option for regenerative medicine and therapeutic applications [13, 14].

This study aims to investigate the efficacy and safety of the topical application of WJ-MSC-derived exosomes in patients with chronic DFUs, thereby exploring a potential new treatment paradigm for this debilitating condition. The outcomes of this research could not only enhance healing rates but also significantly improve the quality of life for individuals suffering from chronic diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:1. Adults aged 18 years or older with type 1 or type 2 diabetes.

2. Presence of a chronic DFU persisting for more than six weeks or showing less than 30% reduction in size after a seven-day standard of care (SOC) management.

3. Ulcers located on the plantar, medial, or lateral aspects of the foot with a size <30 cm².

4. Patients with neuropathic, ischemic, or mixed neuropathic-ischemic ulcers. 5. Revascularization performed for ischemic ulcers before enrollment.

-

Exclusion Criteria:1. Pregnancy or breastfeeding. 2. Presence of venous ulcers or active infections. 3. Exposure of bone, ligaments, or tendons.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2024-04-06 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
Ulcer healing | 20 week
  measuring the percent of wound closure compared to the baseline

CONTACTS AND LOCATIONS:
Locations (1):
- kafr elshaikh university Hospital, Kafrelsheikh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
iam not sure i will share patient private data untill i have aprovement from them